CLINICAL TRIAL: NCT02585037
Title: Changes in Grip Strength by Using Bandage Kinesio Taping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mogi das Cruzes (Other)
Responsible Party: Principal Investigator, Silvia Regina M. S. Boschi, PhD, University of Mogi das Cruzes
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 17119213.0.0000.5497
Record Dates: First submitted 2015-10-20; First posted 2015-10-23 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Hand Strength

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Kinesio Taping for facilitation (Experimental): To provide the facilitation of muscle activity (G1 group) a Kinesio Taping® bandage will be applied to the muscle starting at its origin up to the location of muscle insertion. Bandage in group G1 will be applied following the protocol proposed by method of technical, which defined the direction of the bandage and an applied tension of 10% to 15% (paper off). With a dynamometer Jamar® pressure the grip strength will be messure in four stages: immediately before placing the Kinesio Taping®, 24 h, 48 h, and 72 h after its application.
  Interventions: Other: Kinesio Taping® bandage; Other: Dynamometer Jamar® pressure
- Kinesio Taping for inhibition (Experimental): For inhibition of muscle activity (G2 group), the Kinesio Taping® bandage will be placed over the muscle starting at the insertion location and ending at the muscle origin. Bandage in group G2 will be applied following the protocol proposed by method of technical, which defined the direction of the bandage and an applied tension of 10% to 15% (paper off). With a dynamometer Jamar® pressure the grip strength will be messure in four stages: immediately before placing the Kinesio Taping®, 24 h, 48 h, and 72 h after its application.
  Interventions: Other: Kinesio Taping® bandage; Other: Dynamometer Jamar® pressure
- Kinesio Taping and Placebo (Placebo Comparator): For the control group (G3 group) the Kinesio Taping® bandage will be placed from the lateral extremity to the medial axis. Bandages in the G3 group will be applied laterally to produce a similar visual effect, which control for the placebo effect, but without tension so that a muscle stimulus will be not generated. With a dynamometer Jamar® pressure the grip strength will be messure in four stages: immediately before placing the Kinesio Taping®, 24 h, 48 h, and 72 h after its application.
  Interventions: Other: Dynamometer Jamar® pressure; Other: Placebo

INTERVENTIONS:
Other: Kinesio Taping® bandage — The Kinesio Taping® bandage will be applied in an "I" format in the wrist flexor muscles of a dominant and non-dominant limb in G1 and G2 groups.
  Arms: Kinesio Taping for facilitation; Kinesio Taping for inhibition
Other: Dynamometer Jamar® pressure — The Jamar® dynamometer will be adjusted to the second position for measurement of maximal voluntary strength of handgrip. A muscle contraction period of three seconds will be performed in order to record handgrip strength.
Other: Placebo — For the control group (G3) the Kinesio Taping® bandage will be placed from the lateral extremity to the medial axis.
  Arms: Kinesio Taping and Placebo

SUMMARY:
The Kinesio Taping® method, therapeutic bandage, is another feature can be used in physical therapy, aiming to muscle enhancement, weakened muscles correction, analgesia, among others, by cutaneous stimulation of mechanoreceptors. This study aims to evaluate the efficiency of the use and effects offered by Kinesio Taping® method, changes in muscle strength of grip in normal subjects for clinical application.

DETAILED DESCRIPTION:
A sample of 45 subjects will be divided randomly into three groups (G1: muscle activation technique; G2: muscle inhibition technique; G3: Placebo Effect) aged over 18 years male or female, where it will be initially measured the strength of grip with a dynamometer Jamar® pressure. Then the Kinesio Taping® bandage will be applied in an "I" format in the wrist flexor muscles of a dominant and non-dominant limb in G1, G2, and G3 groups. Investigators will follow the application protocol suggested by method of technical. To provide the facilitation of muscle activity (G1 group) a Kinesio Taping® bandage will be applied to the muscle starting at its origin up to the location of muscle insertion. For inhibition of muscle activity (G2 group), the bandage will be placed over the muscle starting at the insertion location and ending at the muscle origin. For the control group (G3 group) the bandage will be placed from the lateral extremity to the medial axis. The measurement of grip strength was carried out in four stages: immediately before placing the Kinesio Taping®, 24 h, 48 h, and 72 h after its application. After collecting the data statistical Investigators will held the analysis of the data.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged greater than 18 years and with muscle / nerve integrity of upper limbs, hearing and responsive to verbal commands with understanding the information that aware and according to the study.

Exclusion Criteria:

* Individuals who refused to participate in this research and / or do not meet the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change handgrip strength at 72 hours | 24, 48 and 72 hours
  At each stage (24, 48 and 72 hours) the volunteer must perform the measurement of strength three times respecting a period of rest between measurements than a minute.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia R. Boschi, PhD, Principal Investigator — University of Mogi das Cruzes